CLINICAL TRIAL: NCT03866902
Title: Healthy Mothers-Healthy Children: An Intervention With Hispanic Mothers and Their Young Children
Brief Title: Healthy Mothers-Healthy Children Nutrition
Acronym: HMHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hudson Santos, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220623; 1R01NR017199-01 (NIH); 17-0979 (Other: UNC Chapel Hill)
Record Dates: First submitted 2019-02-24; First posted 2019-03-07 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity; Adiposity; Nutrient; Excess; Physical Activity
Keywords: overweight; obesity; adiposity; nutrition; physical activity; Hispanic
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled repeated measures study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The statistician has created a randomization table in RedCap. After enrollment and baseline assessment, dyads will be randomized to either the intervention or control group using a computer-generated randomization table, stratifying by BMI group, overweight (25 - 29.9 kg/m²) and obese (>30 kg/m²), and utilizing blocking to help ensure balance between the groups. Mothers will be informed of their group assignment by telephone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition and Physical Activity Intervention (Experimental): Classes for the intervention mothers will be run by a bilingual interventionist and will last 105 minutes weekly for 12 weeks and then monthly for 6 months.
  Classes for intervention group children will be 105 minutes weekly for 12 weeks and then monthly for 6 months.
  Interventions: Behavioral: Nutrition and Physical Activity Intervention
- English for Second Language Intervention (Active Comparator): Mothers in the control group will receive English as a Second Language (ESL) classes taught by professional ESL teachers; they will receive the same number of contacts and time as the intervention group mothers for 105 minutes weekly for 12 weeks and 105 minutes monthly for 6 months.
  Children in the control group will be read to and color with crayons 105 minutes weekly for 12 weeks and then 105 minutes monthly for 6 months.
  Interventions: Other: English for Second Language Intervention

INTERVENTIONS:
Behavioral: Nutrition and Physical Activity Intervention — Mothers. Twelve weekly classes for one hour focused on nutrition and exercise education and coping skills training followed by a forty five minute exercise class for mothers. Then they will return for one hour for continued support and a forty-five minute exercise class.
  Children. Twelve weekly classes for one hour focused on Color Me Healthy and one hour of free play. Then 6 monthly continued support classes where a Color Me Healthy class will be reviewed and they will have one hour of free play.
  Arms: Nutrition and Physical Activity Intervention
Other: English for Second Language Intervention — Mothers. Control group mothers will receive 12 weekly English for Second Language classes for one hour and forty-five minutes. Then 6 monthly one hour and forty minute follow-up classes receiving English for Second Language material.
  Children. Control group children will receive 12 weekly one hour and forty five minutes of having books read to them. Followed by 6 monthly meetings for one hour and 45 minutes being read to and coloring with crayons.
  Arms: English for Second Language Intervention

SUMMARY:
Using a randomized two-group, repeated measures experimental design, the goal of the proposed study is to investigate the efficacy of a 12-week nutrition and exercise education, physical activity, coping skills training, and home-based physical activity intervention in Hispanic women and their 3-5 year old children and 6 months of continued monthly contact to help overweight and obese Hispanic mothers improve adiposity, weight, health behaviors, and self-efficacy and their 3-5 year old children improve their adiposity and weight gain trajectory and health behaviors.

DETAILED DESCRIPTION:
Hispanic women and children who become overweight or obese are at risk for developing prediabetes, type 2 diabetes, and cardiovascular disease later in life. To date, there have been no interdisciplinary interventions that have targeted Hispanic women and their 3-5 year old children to improve nutrition and physical activity behaviors to manage adiposity and weight in mothers and prevent excessive adiposity and weight gain trajectory in their children. Using a randomized two-group, repeated measures experimental design, the goal of the proposed study is to investigate the efficacy of a 12-week nutrition and exercise education, physical activity, coping skills training, and home-based physical activity intervention in Hispanic women and their 3-5 year old children and 6 months of continued monthly contact to help overweight and obese Hispanic mothers improve adiposity, weight, health behaviors (nutrition and physical activity), and self-efficacy and their 3-5 year old children improve their adiposity and weight gain trajectory and health behaviors (nutrition and physical activity). The investigators will partner with two federally qualified health departments in Durham and Chatham, North Carolina to enroll Hispanic women and their 3-5 year old children and the investigators will partner with community centers to deliver the intervention. A total of 294 Hispanic women with a BMI >25 kg/m² and 294 Hispanic 3-5 year old children with a BMI percentile > 25 will be enrolled over 4 years and randomized to the experimental or equal attention control group. Data will be collected at Time 1 (0 months [baseline]) to Time 2 (9 months [completion of the intervention]) and Time 1 to Time 3 (15 months [after 6 months with no contact from the study staff]). Data collected will include adiposity (primary outcomes: waist circumference, triceps and subscapular skinfolds) in mothers and children and weight (primary outcomes: body mass index [BMI] in mothers and BMI percentile in the children). Secondary outcomes will include health behaviors and self-efficacy in the mothers (Adult Health Behavior Questionnaire, Lifestyle Health Promoting Profile II, 3 day 24-Hour Food Recall, and 7 day Accelerometer, Eating Self-Efficacy Scale and Exercise Self-Efficacy Scale) and in the children (7 day Accelerometer and 3 day 24-Hour Food Recall). The investigators will also evaluate the cost of delivering the program for public health departments. Data analysis will use general linear mixed models to test the hypotheses. Decreasing overweight and obesity in Hispanic women and slowing adiposity and weight gain trajectory in young Hispanic children is urgently needed to decrease morbidity, mortality, and future health care costs. The knowledge to be gained from this study may provide a foundation for extending this intervention to other Hispanic mothers and children in other communities to assist mothers in managing their weight and preventing excessive adiposity and weight gain in their children. This approach is translatable, real-world, and could be replicated in other areas of the United States.

ELIGIBILITY:
Inclusion criteria for mothers will be:

* age 18 years or older
* self-identification as Hispanic
* limited English proficiency; little acculturation, as measured by the Short Acculturation Scale for Hispanics with a score from 1.00 to 2.99
* ability to understand spoken Spanish
* a BMI >25kg/m^2
* residence with the child
* consent to join the study and consent for their child to join the study.

Inclusion criteria for children will be:

* age 3-5 years
* ability to understand spoken Spanish
* a BMI > 25th percentile for age and gender

Exclusion criteria for mothers will be:

* heart murmur
* congenital heart disease
* family history of sudden death
* difficulty exercising
* psychological problems

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 578 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hudson Santos, PhD, Principal Investigator — University of Miami
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry DC, Gonzales C, Montano NP, Perreira KM, Ammerman AS, Crandell J, Evenson KR, Faith MS, Waters H, Linares C, Comicronrtes YI, Perrin EM. Rationale, design, and methodology for the healthy mothers-healthy children study: a randomized controlled trial. BMC Nutr. 2019 Dec 16;5:58. doi: 10.1186/s40795-019-0322-7. eCollection 2019. PMID 32153971

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Dyad study design. Only one consent was signed by mother to agree to both mother and child to participant in the study; therefore, a total of 578 were enrolled in the study. 4 signed the consent but were not randomized into the groups for this study and did not participate in the intervention because of a lack of desire to participate just prior to the intervention starting; therefore, were not enrolled in the arms. Mother/child dyads that went into the arms/groups Total= 574.
Groups:
- Nutrition and Physical Activity Intervention: Classes for the intervention mothers will be run by a bilingual interventionist and will last 105 minutes weekly for 12 weeks and then monthly for 6 months.
  Classes for intervention group children will be 105 minutes weekly for 12 weeks and then monthly for 6 months.
  Nutrition and Physical Activity Intervention: Mothers. Twelve weekly classes for one hour focused on nutrition and exercise education and coping skills training followed by a forty five minute exercise class for mothers. Then they will return for one hour for continued support and a forty-five minute exercise class.
  Children. Twelve weekly classes for one hour focused on Color Me Healthy and one hour of free play. Then 6 monthly continued support classes where a Color Me Healthy class will be reviewed and they will have one hour of free play.
- English for Second Language Intervention: Mothers in the control group will receive English as a Second Language (ESL) classes taught by professional ESL teachers; they will receive the same number of contacts and time as the intervention group mothers for 105 minutes weekly for 12 weeks and 105 minutes monthly for 6 months.
  Children in the control group will be read to and color with crayons 105 minutes weekly for 12 weeks and then 105 minutes monthly for 6 months.
  English for Second Language Intervention: Mothers. Control group mothers will receive 12 weekly English for Second Language classes for one hour and forty-five minutes. Then 6 monthly one hour and forty minute follow-up classes receiving English for Second Language material.
  Children. Control group children will receive 12 weekly one hour and forty five minutes of having books read to them. Followed by 6 monthly meetings for one hour and 45 minutes being read to and coloring with crayons.
Period: Overall Study
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Started | 288 | 286
Mother | 144 | 143
Child | 144 | 143
Completed | 172 | 180
Not Completed | 116 | 106
Not completed — Lost to Follow-up | 98 | 82
Not completed — Pregnancy | 18 | 24

BASELINE CHARACTERISTICS:
Population: This is a dyad study. Data was collected for both mother and child for the gender and age category. Ethnicity was only collected for mother.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention | Total
Number analyzed (Participants) | 288 | 286 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One of the mother's data for age was not collected.
  years
    Mother: number analyzed (Participants) | 144 | 142 | 286
    Mother | 34.9 (6.63) | 34.6 (6.60) | 34.8 (6.60)
    Child: number analyzed (Participants) | 144 | 143 | 287
    Child | 4.33 (0.988) | 4.42 (0.905) | 4.38 (0.947)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One of the child's data for the sex was not collected.
  Participants
    Mother: number analyzed (Participants) | 144 | 143 | 287
    Mother: Female | 144 | 143 | 287
    Mother: Male | 0 | 0 | 0
    Child: number analyzed (Participants) | 144 | 142 | 286
    Child: Female | 77 | 75 | 152
    Child: Male | 67 | 67 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only data for the mother was collected.
  Participants
    number analyzed (Participants) | 144 | 143 | 287
    Hispanic or Latino | 144 | 143 | 287
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mother's Height From Baseline (Time 1) to Time 2
Description: Height in centimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | -0.00977 (0.485) | 0.000505 (0.00503)

2. Primary Outcome: Change in Mother's Height From Baseline (Time 1) to Time 3
Description: Height in centimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | -0.00116 (0.0108) | 0 (0)

3. Primary Outcome: Change in Children's Height From Baseline (Time 1) to Time 2
Description: Height in centimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | 8.62 (3.38) | 7.86 (3.20)

4. Primary Outcome: Change in Children's Height From Baseline (Time 1) to Time 3
Description: Height in centimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | 11.5 (3.39) | 10.7 (3.65)

5. Primary Outcome: Change in Mother's Weight From Baseline (Time 1) to Time 2
Description: Weight in kilograms
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Kilograms | 0.0776 (3.68) | -0.431 (4.08)

6. Primary Outcome: Change in Mother's Weight From Baseline (Time 1) to Time 3
Description: Weight in kilograms
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Kilograms | 0.488 (4.25) | 0.435 (4.24)

7. Primary Outcome: Change in Children's Weight From Baseline (Time 1) to Time 2
Description: Weight in kilograms
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Kilograms | 3.36 (2.50) | 3.11 (2.40)

8. Primary Outcome: Change in Children's Weight From Baseline (Time 1) to Time 3
Description: Weight in kilograms
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Kilograms | 4.81 (3.39) | 4.63 (3.33)

9. Primary Outcome: Change in Mother's BMI From Baseline (Time 1) to Time 2
Description: Calculation of BMI in Mothers in kilograms divided by meters squared
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
kg/m^2 | 0.0437 (1.62) | -0.170 (1.66)

10. Primary Outcome: Change in Mother's BMI From Baseline (Time 1) to Time 3
Description: Calculation of BMI in Mothers in kilograms divided by meters squared
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
kg/m^2 | 0.194 (1.86) | 0.195 (1.73)

11. Primary Outcome: Change in Children's BMI Percentile From Baseline (Time 1) to Time 2
Description: Calculation of BMI measured in percentage in Children. Calculated by the percentage of the mean BMI.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: percentage of children's BMI
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
percentage of children's BMI | -7.21 (18.8) | -7.69 (18.9)

12. Primary Outcome: Change in Children's BMI Percentile From Baseline (Time 1) to Time 3
Description: Calculation of BMI Percentile in Children. Calculated by the percentage of the mean BMI.
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: percentage of children's BMI
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
percentage of children's BMI | -8.69 (18.8) | -7.21 (20.8)

13. Primary Outcome: Change in Mother's Adiposity (Waist Circumference) From Baseline (Time 1) to Time 2
Description: Waist Circumference in centimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | 0.172 (5.42) | 0.661 (4.62)

14. Primary Outcome: Change in Mother's Adiposity (Waist Circumference) From Baseline (Time 1) to Time 3
Description: Waist Circumference in centimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | 0.769 (6.77) | 0.399 (6.93)

15. Primary Outcome: Change in Children's Adiposity (Waist Circumference) From Baseline (Time 1) to Time 2
Description: Waist circumference in centimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | 4.38 (4.74) | 4.77 (4.70)

16. Primary Outcome: Change in Children's Adiposity (Waist Circumference) From Baseline (Time 1) to Time 3
Description: Waist circumference in Centimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Centimeters | 5.00 (4.61) | 5.71 (5.67)

17. Primary Outcome: Change in Mother's Adiposity (Triceps Skinfold) From Baseline (Time 1) to Time 2
Description: Triceps skinfolds in Millimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | -0.421 (6.85) | -0.848 (7.16)

18. Primary Outcome: Change in Mother's Adiposity (Triceps Skinfold) From Baseline (Time 1) to Time 3
Description: Triceps skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | -1.77 (6.95) | -0.854 (7.42)

19. Primary Outcome: Change in Children's Adiposity (Triceps Skinfold) From Baseline (Time 1) to Time 2
Description: Triceps skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | 0.734 (4.51) | 0.920 (5.31)

20. Primary Outcome: Change in Children's Adiposity (Triceps Skinfold) From Baseline (Time 1) to Time 3
Description: Triceps skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | 1.02 (4.60) | 1.35 (4.45)

21. Primary Outcome: Change in Mother's Adiposity (Subscapular Skinfolds) Baseline (Time 1) to Time 2
Description: Subscapular skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | 0.697 (5.98) | 0.558 (6.64)

22. Primary Outcome: Change in Mother's Adiposity (Subscapular Skinfolds) Baseline (Time 1) to Time 3
Description: Subscapular skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | 1.00 (6.14) | 0.737 (7.17)

23. Primary Outcome: Change in Children's Adiposity (Subscapular Skinfolds) From Baseline (Time 1) to Time 2
Description: Subscapular skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | 1.13 (3.40) | 0.984 (3.89)

24. Primary Outcome: Change in Children's Adiposity (Subscapular Skinfolds) Baseline (Time 1) to Time 3
Description: Subscapular skinfolds in millimeters
Time Frame: Baseline (Time 1), Time 3 (approximately 15 months)
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Nutrition and Physical Activity Intervention | English for Second Language Intervention
Number analyzed (Participants) | 144 | 143
Millimeters | 1.06 (3.79) | 1.36 (4.42)

25. Secondary Outcome: Change in Health Behaviors (Adult Health Behavior Questionnaire) in Mothers Baseline (Time 1) to Time 2
Description: There are 23 questions with a range of answers for each question. Each question is scored individually as a predetermined healthy or unhealthy choice.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

26. Secondary Outcome: Change in Health Behaviors (Adult Health Behavior Questionnaire) in Mothers Baseline (Time 1) to Time 3
Description: as for outcome 25
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

27. Secondary Outcome: Change in Health Behaviors (Health Promoting Lifestyle Profile II) in Mothers Baseline (Time 1) to Time 2
Description: There are 34 questions and the answer choices are never, sometime, often or routinely. Never is scored a 0, sometimes is scored a 1, often is scored a 2 and routine is scored a 3. The 34 questions are summed to provide a total score. A higher score reflects healthier behaviors and a lower score reflects unhealthier behaviors.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

28. Secondary Outcome: Change in Health Behaviors (Health Promoting Lifestyle Profile II) in Mothers From Baseline (Time 1) to Time 3
Description: as for outcome 27
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

29. Secondary Outcome: Change in Health Behaviors (24 Hour Food Recall) for 3 Days in Mothers From Baseline (Time 1) to Time 2
Description: Phone Interview with the Mother on a Monday, Tuesday and Wednesday. The research assistant will ask the mother what she ate at breakfast, lunch, dinner and snacks and approximate amounts. This information will be entered into nutritionistpro a software program. Then total calories, protein, carbohydrate and fat can be calculated for each day.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

30. Secondary Outcome: Change in Health Behaviors (24 Hour Food Recall) for 3 Days in Mothers From Baseline (Time 1) to Time 3
Description: as for outcome 29
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

31. Secondary Outcome: Change in Health Behaviors (24 Hour Food Recall) for 3 Days in Children From Baseline (Time 1) to Time 2
Description: Phone Interview with the Mother on a Monday, Tuesday and Wednesday. The research assistant will ask the mother what her child ate at breakfast, lunch, dinner and snacks and approximate amounts. This information will be entered into nutritionistpro a software program. Then total calories, protein, carbohydrate and fat can be calculated for each day.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

32. Secondary Outcome: Change in Health Behaviors (24 Hour Food Recall) for 3 Days in Children From Baseline (Time 1) to Time 3
Description: as for outcome 31
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

33. Secondary Outcome: Change in Health Behaviors (Accelerometer Measurement for 7 Days) in Mothers From Baseline (Time 1) to Time 2
Description: The Mother will wear an accelerometer for 7 days total. This information will be uploaded into the computer to provide data on low, moderate, and high intensity physical activity.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

34. Secondary Outcome: Change in Health Behaviors (Accelerometer Measurement for 7 Days) in Mothers From Baseline (Time 1) to Time 3
Description: as for outcome 33
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

35. Secondary Outcome: Change in Health Behaviors (Accelerometer Measurement for 7 Days) in Children From Baseline (Time 1) to Time 2
Description: The Child will wear an accelerometer for 7 days total. This information will be uploaded into the computer to provide data on low, moderate, and high intensity physical activity.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

36. Secondary Outcome: Change in Health Behaviors (Accelerometer Measurement for 7 Days) in Children From Baseline (Time 1) to Time 3
Description: as for outcome 35
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

37. Secondary Outcome: Change in Eating Self-Efficacy Questionnaire in Mothers From Baseline (Time 1) to Time 2
Description: This is a 25 question questionnaire asking how much difficulty the Mother has with controlling her eating in social situations and everyday. The range of scores go from 1 to 7 with 1 being no difficulty controlling eating to 4 moderate difficulty controlling eating to 7 the most difficulty controlling eating. The 25 questions are added to produce a total score. A lower score equals less difficulty controlling eating and a higher score equals more difficulty controlling eating.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

38. Secondary Outcome: Change in Eating Self-Efficacy Questionnaire in Mothers From Baseline (Time 1) to Time 3
Description: as for outcome 37
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

39. Secondary Outcome: Change in Exercise Self-Efficacy Questionnaire in Mothers From Baseline (Time 1) to Time 2
Description: This is a 18 question questionnaire asking how much difficulty the Mother has with exercise. The range of scores go from 1 to 10 with 1 being she can not do it at all and 6 that she can moderately do exercise and a 10 that she is certain she can do it. The numbers are summed for a total score. A lower number indicates that the mother has a lot of difficulty exercising and a higher number means that the mother is more certain she can exercise.
Time Frame: Baseline (Time 1), Time 2 (Intervention completion, approximately 9 months)
Reporting Status: Not Posted

40. Secondary Outcome: Change in Exercise Self-Efficacy Questionnaire in Mothers From Baseline (Time 1) to Time 3
Description: as for outcome 39
Time Frame: Baseline (Time 1), Time 3 (after 6 months with no contact from the study staff, approximately 15 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months
Description: Both the mother and child were monitored for 4 years for the duration over which adverse events were monitored/assessed
Groups:
- Nutrition and Physical Activity Intervention-Mother: Classes for the intervention mothers will be run by a bilingual interventionist and will last 105 minutes weekly for 12 weeks and then monthly for 6 months.
- English for Second Language Intervention-Mother: Mothers in the control group will receive English as a Second Language (ESL) classes taught by professional ESL teachers; they will receive the same number of contacts and time as the intervention group mothers for 105 minutes weekly for 12 weeks and 105 minutes monthly for 6 months.
- Nutrition and Physical Activity Intervention-Child: Classes for intervention group children will be 105 minutes weekly for 12 weeks and then monthly for 6 months.
- English for Second Language Intervention-Child: Children in the control group will be read to and color with crayons 105 minutes weekly for 12 weeks and then 105 minutes monthly for 6 months.
Arm/Group | Nutrition and Physical Activity Intervention-Mother | English for Second Language Intervention-Mother | Nutrition and Physical Activity Intervention-Child | English for Second Language Intervention-Child
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/143 | 0/144 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/143 | 0/144 | 0/143
Other Adverse Events (participants affected / at risk) | 0/144 | 0/143 | 0/144 | 0/143

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03866902/Prot_SAP_000.pdf